CLINICAL TRIAL: NCT00680745
Title: A 24-Week,Int.,Rand.,Double-blind,Parallel-group,Multi-centre, Plac.-Controlled Phase III Study With a 24-Wk Ext.Per.to Eval.the Efficacy and Safety of Dapagliflozin in Comb.With Glimepiride (a Sulphonylurea) in Subjects With Type2 Diab.Who Have Inadeq. Glycaemic Control on Glimepiride Therapy Alone
Brief Title: Efficacy and Safety of Dapagliflozin in Combination With Glimepiride (a Sulphonylurea) in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1690C00005
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes
Keywords: Dapagliflozin; efficacy; safety; sulphonylurea; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; glimepiride; Metformin; Pioglitazone; Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): dapagliflozin 2.5mg + Glimepiride
  Interventions: Drug: dapagliflozin; Drug: Glimepiride; Drug: metformin hydrochloride; Drug: pioglitazone hydrochloride; Drug: Rosiglitazone
- 2 (Experimental): dapagliflozin 5mg + Glimepiride
  Interventions: Drug: dapagliflozin; Drug: Glimepiride; Drug: metformin hydrochloride; Drug: pioglitazone hydrochloride; Drug: Rosiglitazone
- 3 (Experimental): dapagliflozin 10mg + Glimepiride
  Interventions: Drug: dapagliflozin; Drug: Glimepiride; Drug: metformin hydrochloride; Drug: pioglitazone hydrochloride; Drug: Rosiglitazone
- 4 (Placebo Comparator): Placebo + Glimepiride
  Interventions: Drug: Glimepiride; Drug: metformin hydrochloride; Drug: pioglitazone hydrochloride; Drug: Rosiglitazone

INTERVENTIONS:
Drug: dapagliflozin — tablet oral 2.5, 5, or 10 mg total daily dose once daily 48 weeks
  Arms: 1; 2; 3
Drug: Glimepiride — tablet oral 2.5, 5, or 10 mg total daily dose once daily 48 weeks
  Other Names: Amaryl
Drug: metformin hydrochloride — rescue medication oral dosing in accordance with the manufacturer's recommendations and clinical practice
  Other Names: Glucophage
Drug: pioglitazone hydrochloride — rescue medication oral dosing in accordance with the manufacturer's recommendations and clinical practice
  Other Names: Actos
Drug: Rosiglitazone — rescue medication oral dosing in accordance with the manufacturer's recommendations and clinical practice
  Other Names: Avandia

SUMMARY:
This study is being carried out to see if dapagliflozin in addition to glimepiride (sulphonylurea) is effective and safe in treating patients with type 2 diabetes when compared to glimepiride alone.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Treatment with a stable sulphonylurea monotherapy dose that is at least half the maximal recommended dose for a minimum of 8 weeks prior to study
* Inadequate glycaemic control, defined as A1C ≥ 7.0 % and ≤ 10%

Exclusion Criteria:

* Type 1 Diabetes
* Hepatic (liver) impairment
* Renal (kidney) failure or dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Strojek, Prof. Dr., Principal Investigator — Silesian Medical University3-Maja 13/15, 41-800 Zabrze; Poland
Locations (66):
- Czechia (10):
  - Research Site, Blansko
  - Research Site, Bruntál
  - Research Site, Břeclav
  - Research Site, Hodonín
  - Research Site, Ostrava - Belsky Les
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Pribram VIII
  - Research Site, Rakovník
  - Research Site, Semily
- Hungary (14):
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Csongrád
  - Research Site, Eger
  - Research Site, Gyöngyös
  - Research Site, Kecskemét
  - Research Site, Makó
  - Research Site, Miskolc
  - Research Site, Mosonmagyaróvár
  - Research Site, Siófok
  - Research Site, Szentes
  - Research Site, Tát
  - Research Site, Zalaegerszeg
- Philippines (4):
  - Research Site, Cebu City
  - Research Site, Manila
  - Research Site, Marikina City
  - Research Site, Pasig
- Poland (22):
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Chojnice
  - Research Site, Chrzanów
  - Research Site, Ciechocinek
  - Research Site, Czechowice-Dziedzice
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Gniewkowo
  - Research Site, Grudziądz
  - Research Site, Iława
  - Research Site, Krakow
  - Research Site, Mrągowo
  - Research Site, Poznan
  - Research Site, Płock
  - Research Site, Ruda Śląska
  - Research Site, Sopot
  - Research Site, Torun
  - Research Site, Wroclaw
  - Research Site, Zabrze
  - Research Site, Zielona Góra
  - Research Site, Żory
- South Korea (8):
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Suwon, Gyeonggi-do
  - Research Site, Jeonju, Jeollabuk-do
  - Research Site, Bucheon-si
  - Research Site, Incheon
  - Research Site, Seongnam
  - Research Site, Seoul
  - Research Site, Uljeongbu
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
- Ukraine (6):
  - Research Site, Dnipropetrov'sk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya

REFERENCES:
- [Derived] Shah M, Stolbov L, Yakovleva T, Tang W, Sokolov V, Penland RC, Boulton D, Parkinson J. A model-based approach to investigating the relationship between glucose-insulin dynamics and dapagliflozin treatment effect in patients with type 2 diabetes. Diabetes Obes Metab. 2021 Apr;23(4):991-1000. doi: 10.1111/dom.14305. Epub 2021 Jan 25. PMID 33368935
- [Derived] Strojek K, Yoon KH, Hruba V, Elze M, Langkilde AM, Parikh S. [Effect of dapagliflozin in patients with type 2 diabetes who have inadequate glycaemic control with glimepiride]. Dtsch Med Wochenschr. 2013 Apr;138 Suppl 1:S16-26. doi: 10.1055/s-0032-1305277. Epub 2013 Mar 25. German. PMID 23529567
- [Derived] Strojek K, Yoon KH, Hruba V, Elze M, Langkilde AM, Parikh S. Effect of dapagliflozin in patients with type 2 diabetes who have inadequate glycaemic control with glimepiride: a randomized, 24-week, double-blind, placebo-controlled trial. Diabetes Obes Metab. 2011 Oct;13(10):928-38. doi: 10.1111/j.1463-1326.2011.01434.x. PMID 21672123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment: 859 (597 randomized and 592 in the Full Analysis Set) Study Start Date:April 2008 Study Completion Date:May 2010 Primary Completion Date: November 2009 (Final data collection date for primary outcome measure)
Pre-assignment Details: Reasons for enrolled participants not being randomised: 229 incorrect enrollment, 4 adverse event, 23 withdrew consent, 2 lost to follow up and 4 other.
Groups:
- Dapagliflozin 2.5mg + Glimepiride: Dapagliflozin tablet 2.5 mg once daily plus glimepiride
- Dapagliflozin 5mg + Glimepiride: Dapagliflozin tablet 5 mg once daily plus glimepiride
- Dapagliflozin 10mg + Glimepiride: Dapagliflozin tablet 10 mg once daily plus glimepiride
- Placebo + Glimepiride: Placebo comparator plus glimepiride
Period: Overall Study
Arm/Group | Dapagliflozin 2.5mg + Glimepiride | Dapagliflozin 5mg + Glimepiride | Dapagliflozin 10mg + Glimepiride | Placebo + Glimepiride
Started | 154 (Safety Analysis Set) | 145 (Safety Analysis Set) | 151 (Safety Analysis Set) | 146 (Safety Analysis Set)
Completed | 140 | 132 | 141 | 133
Not Completed | 14 | 13 | 10 | 13
Not completed — Withdrawal by Subject | 8 | 3 | 2 | 8
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Death | 1 | 0 | 1 | 0
Not completed — Adverse Event | 5 | 3 | 3 | 3
Not completed — Poor/Non-compliance | 0 | 3 | 0 | 0
Not completed — Subject No Longer Meets Study Criteria | 0 | 2 | 0 | 2
Not completed — False Treatment | 0 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set defined as all randomized participants (as randomized) who received at least one dose of double-blind study medication, who have a non-missing baseline value and at least one post-baseline efficacy value for at least one efficacy variable during double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 2.5mg + Glimepiride | Dapagliflozin 5mg + Glimepiride | Dapagliflozin 10mg + Glimepiride | Placebo + Glimepiride | Total
Number analyzed (Participants) | 154 | 142 | 151 | 145 | 592
Age Continuous [Mean (Standard Deviation); unit: years] | 59.9 (10.14) | 60.2 (9.73) | 58.9 (8.32) | 60.3 (10.16) | 59.8 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 71 | 85 | 74 | 307
  Male | 77 | 71 | 66 | 71 | 285
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 108 | 96 | 106 | 101 | 411
  Asian | 46 | 46 | 45 | 44 | 181
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.01 (5.120) | 29.84 (5.182) | 29.75 (5.641) | 29.74 (4.569) | 29.84 (5.135)
HbA1c [Mean (Standard Deviation); unit: Percent] | 8.11 (0.749) | 8.12 (0.781) | 8.07 (0.790) | 8.15 (0.736) | 8.11 (0.763)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in HbA1c Levels
Description: To assess the efficacy of dapagliflozin compared to placebo as add-on therapy to glimepiride in improving glycemic control in participants with type 2 diabetes, as determined by the change in HbA1C levels from baseline to the end of the 24-week double-blind treatment period.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Groups:
- Dapagliflozin 10mg + Glimepiride: Dapagliflozin tablet 2.5 mg once daily plus glimepiride
Arm/Group | Dapagliflozin 2.5mg + Glimepiride | Dapagliflozin 5mg + Glimepiride | Dapagliflozin 10mg + Glimepiride | Placebo + Glimepiride
Number analyzed (Participants) | 154 | 142 | 150 | 143
Percent | -0.58 [-0.69 to -0.46] | -0.63 [-0.75 to -0.50] | -0.82 [-0.94 to -0.70] | -0.13 [-0.26 to -0.01]
Statistical Analysis 1: Comparison: Dapagliflozin 2.5mg + Glimepiride vs Placebo + Glimepiride; The null hypothesis is given as H0: mean(treat) minus mean(placebo) = 0 versus HA: mean(treat) minus mean(placebo) =/= 0 (with alpha = 0.019 applying Dunnett's adjustment, two-sided); Test type: Superiority or Other; p < 0.0001, ANCOVA — significant at alpha=0.019 (2-sided) applying Dunnett's adjustment. A hierarchical closed testing procedure was used to control the Type I error rate across the primary and key secondary endpoints; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.61 to -0.27], Standard Error of Mean 0.0867
Statistical Analysis 2: Comparison: Dapagliflozin 5mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.67 to -0.32], Standard Error of Mean 0.0885
Statistical Analysis 3: Comparison: Dapagliflozin 10mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-0.86 to -0.51], Standard Error of Mean 0.0873

2. Secondary Outcome: Adjusted Mean Change in Body Weight
Description: To show that dapagliflozin plus glimepiride results in greater reduction in body weight or less weight gain after 24 weeks of treatment when compared to placebo plus glimepiride.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Dapagliflozin 2.5mg + Glimepiride | Dapagliflozin 5mg + Glimepiride | Dapagliflozin 10mg + Glimepiride | Placebo + Glimepiride
Number analyzed (Participants) | 154 | 142 | 151 | 145
kg | -1.18 [-1.62 to -0.75] | -1.56 [-2.01 to -1.11] | -2.26 [-2.70 to -1.83] | -0.72 [-1.16 to -0.28]
Statistical Analysis 1: Comparison: Dapagliflozin 2.5mg + Glimepiride vs Placebo + Glimepiride; The null hypothesis is given as H0: mean(treat) minus mean(placebo) = 0 versus HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.1410, ANCOVA — not significant at alpha=0.05 (2-sided). Primary and key secondary endpoints are tested following a hierarchical closed testing procedure within treatment group; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-1.08 to 0.15], Standard Error of Mean 0.3153
Statistical Analysis 2: Comparison: Dapagliflozin 5mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0091, ANCOVA — significant at alpha=0.05 (2-sided). Primary and key secondary endpoints are tested following a hierarchical closed testing procedure within treatment group; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.47 to -0.21], Standard Error of Mean 0.3217
Statistical Analysis 3: Comparison: Dapagliflozin 10mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 2]; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-2.17 to -0.92], Standard Error of Mean 0.3168

3. Secondary Outcome: Adjusted Mean Change in 2-h Post-challenge Plasma Glucose Rise
Description: To show that dapagliflozin plus glimepiride results in greater reductions in the 2-h post-challenge plasma glucose rise as a response to an oral glucose tolerance test (OGTT) from baseline to Week 24.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dapagliflozin 2.5mg + Glimepiride | Dapagliflozin 5mg + Glimepiride | Dapagliflozin 10mg + Glimepiride | Placebo + Glimepiride
Number analyzed (Participants) | 126 | 117 | 132 | 109
mg/dL | -37.5 [-46.7 to -28.3] | -32.0 [-41.5 to -22.5] | -34.9 [-43.8 to -25.9] | -6.0 [-15.8 to 3.9]
Statistical Analysis 1: Comparison: Dapagliflozin 2.5mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANCOVA — Not significant. Hierarchical closed testing procedure within treatment group stopped at previous endpoint; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -31.5, 95% CI 2-sided [-45.0 to -18.0], Standard Error of Mean 6.874
Statistical Analysis 2: Comparison: Dapagliflozin 5mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 2, analysis 2]; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -26.0, 95% CI 2-sided [-39.7 to -12.3], Standard Error of Mean 6.968
Statistical Analysis 3: Comparison: Dapagliflozin 10mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 2]; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -28.9, 95% CI 2-sided [-42.2 to -15.6], Standard Error of Mean 6.770

4. Secondary Outcome: Proportion of Participants Achieving Glycemic Response Defined as HbA1c <7%
Description: To show that dapagliflozin plus glimepiride results in a larger proportion of participants achieving a therapeutic glycemic response, defined as HbA1c < 7% after 24 weeks of treatment, compared to placebo plus glimepiride.
Time Frame: At Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dapagliflozin 2.5mg + Glimepiride | Dapagliflozin 5mg + Glimepiride | Dapagliflozin 10mg + Glimepiride | Placebo + Glimepiride
Number analyzed (Participants) | 154 | 142 | 150 | 143
Percentage of participants | 26.8 [20.2 to 33.3] | 30.3 [23.4 to 37.1] | 31.7 [24.7 to 38.7] | 13.0 [7.6 to 18.4]
Statistical Analysis 1: Comparison: Dapagliflozin 2.5mg + Glimepiride vs Placebo + Glimepiride; H0: proportion(treat) minus proportion(placebo) = 0 versus the alternative HA: proportion(treat) minus proportion(placebo) =/= 0; Test type: Superiority or Other; Regression, Logistic — Not significant. Hierarchical closed testing procedure within treatment group stopped at previous endpoint; Based on methodology of Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu, with adjustment for baseline value; Risk Difference (RD) = 13.7, 95% CI 2-sided [5.4 to 22.1], Standard Error of Mean 4.265
Statistical Analysis 2: Comparison: Dapagliflozin 5mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 2, analysis 2]; Based on methodology of Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu, with adjustment for baseline value; Risk Difference (RD) = 17.3, 95% CI 2-sided [8.7 to 25.9], Standard Error of Mean 4.392
Statistical Analysis 3: Comparison: Dapagliflozin 10mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 2, analysis 2]; Based on methodology of Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu, with adjustment for baseline value; Risk Difference (RD) = 18.7, 95% CI 2-sided [9.9 to 27.4], Standard Error of Mean 4.457

5. Secondary Outcome: Adjusted Mean Change in Body Weight for Participants With Baseline Body Mass Index (BMI)≥27 kg/m2
Description: To show that dapagliflozin plus glimepiride results in greater reductions in body weight or less weight gain in participants with baseline BMI ≥27 kg/m2 after 24 weeks of treatment when compared to placebo plus glimepiride.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with baseline BMI of 27 kg/m2 or more and Week 24 (LOCF) body weight value
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Dapagliflozin 2.5mg + Glimepiride | Dapagliflozin 5mg + Glimepiride | Dapagliflozin 10mg + Glimepiride | Placebo + Glimepiride
Number analyzed (Participants) | 104 | 97 | 99 | 103
kg | -1.17 [-1.75 to -0.59] | -1.74 [-2.34 to -1.15] | -2.47 [-3.06 to -1.88] | -0.80 [-1.38 to -0.22]
Statistical Analysis 1: Comparison: Dapagliflozin 2.5mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANCOVA — Not significant. Hierarchical closed testing procedure within treatment group stopped at previous endpoint; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-1.19 to 0.45], Standard Error of Mean 0.4159
Statistical Analysis 2: Comparison: Dapagliflozin 5mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0262, ANCOVA — [p-value comment as in outcome 2, analysis 2]; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-1.78 to -0.11], Standard Error of Mean 0.4234
Statistical Analysis 3: Comparison: Dapagliflozin 10mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 2]; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -1.67, 98% CI 2-sided [-2.50 to -0.84], Standard Error of Mean 0.4211

6. Secondary Outcome: Adjusted Mean Change in Fasting Plasma Glucose (FPG)
Description: To show that dapagliflozin plus glimepiride leads to greater reductions in FPG after 24 weeks of treatment compared to placebo plus glimepiride.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dapagliflozin 2.5mg + Glimepiride | Dapagliflozin 5mg + Glimepiride | Dapagliflozin 10mg + Glimepiride | Placebo + Glimepiride
Number analyzed (Participants) | 154 | 142 | 150 | 145
mg/dL | -16.8 [-21.7 to -12.0] | -21.2 [-26.3 to -16.2] | -28.5 [-33.4 to -23.6] | -2.0 [-6.9 to 3.0]
Statistical Analysis 1: Comparison: Dapagliflozin 2.5mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANCOVA — Not significant. Hierarchical closed testing procedure within treatment group stopped at previous endpoint; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -14.9, 95% CI 2-sided [-21.8 to -7.9], Standard Error of Mean 3.522
Statistical Analysis 2: Comparison: Dapagliflozin 5mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 2]; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -19.3, 95% CI 2-sided [-26.3 to -12.2], Standard Error of Mean 3.594
Statistical Analysis 3: Comparison: Dapagliflozin 10mg + Glimepiride vs Placebo + Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 2]; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -26.5, 95% CI 2-sided [-33.5 to -19.5], Standard Error of Mean 3.545

ADVERSE EVENTS:
Time Frame: Non-serious/serious adverse events on or after the first day and on or prior to the last day of the 24-week double-blind treatment period plus 4/30 days or up to follow-up visit if earlier, or up to and incl the start date of extension period if earlier.
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Arm/Group | Dapagliflozin 2.5mg + Glimepiride | Dapagliflozin 5mg + Glimepiride | Dapagliflozin 10mg + Glimepiride | Placebo + Glimepiride
Serious Adverse Events (participants affected / at risk) | 11/154 | 10/145 | 9/151 | 7/146
Other Adverse Events (participants affected / at risk) | 22/154 | 19/145 | 18/151 | 15/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin 2.5mg + Glimepiride (N=154) | Dapagliflozin 5mg + Glimepiride (N=145) | Dapagliflozin 10mg + Glimepiride (N=151) | Placebo + Glimepiride (N=146)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 1 | 1 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0 | 0 | 0
AORTIC VALVE DISEASE MIXED (Cardiac disorders) | 0 | 0 | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 0 | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 0 | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1 | 0 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 0 | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
GASTRODUODENITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0
MULTIPLE ALLERGIES (Immune system disorders) | 1 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 2 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
OBESITY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
RECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0 | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 0 | 0 | 1 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin 2.5mg + Glimepiride (N=154) | Dapagliflozin 5mg + Glimepiride (N=145) | Dapagliflozin 10mg + Glimepiride (N=151) | Placebo + Glimepiride (N=146)
NASOPHARYNGITIS (Infections and infestations) | 3 | 8 | 5 | 4
HYPERTENSION (Vascular disorders) | 8 | 2 | 2 | 6
Hypoglycemia (Endocrine disorders) | 11 | 10 | 12 | 7

LIMITATIONS AND CAVEATS:
For participants who did not complete 24 weeks LOCF (last observation carried forward) was used. Only values prior to rescue medication were used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.